CLINICAL TRIAL: NCT04338646
Title: Is the Severity of Urinary Disorders Related to Falls in People With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gérard Amarenco (Other)
Responsible Party: Sponsor-Investigator, Gérard Amarenco, Head of Neuro-Urology department, Tenon Hospital, Pierre and Marie Curie University
Organization: Pierre and Marie Curie University (Other)
Other Study IDs: GREEN GRC01 P
Record Dates: First submitted 2020-04-04; First posted 2020-04-08 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Fall; Multiple Sclerosis; Lower Urinary Tract Symptoms
Keywords: Fall; multiple sclerosis; lower urinary tract symptoms; overactive bladder
MeSH Terms: conditions — Multiple Sclerosis; Lower Urinary Tract Symptoms; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled: Patient with multiple sclerosis and lower urinary tract symptoms, age >18 Expanded Disability Status Scale score between 1 and 6.5
  Interventions: Other: Clinical tests

INTERVENTIONS:
Other: Clinical tests — Questionnaire about urinary symptoms, gait difficulties, fear of falling. Clinical test: Time to be Ready to Void

SUMMARY:
Falls are a common problem in people with multiple sclerosis (PwMS) and can lead to severe consequences (trauma, fear of falling, reduction of social activities). Prevention of falls is one of the priority targets of rehabilitation for PwMS and walking difficulties, which can result of different factors (motor impairment, ataxia, sensitive disorders, fatigability…). Urinary incontinence has been evoked as predictive of falls. But lower urinary tract symptoms (LUTSs) are frequent in PwMS, the prevalence of LUTSs is high (32-96.8%) and increases with MS duration and severity of neurological deficiencies and disabilities. Overactive bladder (OAB) is the most common symptom. Despite its high prevalence and impact on quality of life, the severity of LUTSs has never been studied as specific risk factor of falling. However, urinary urgency and urinary incontinence could lead to precipitation and thus could increase the risk of falling in these patients.

The aim of the study was to assess the relationship between severity of LUTSs and risk of falling in PwMS.

Patients were asked about the number of falls in the past three months and in the past year, and the circumstances in which they occurred (frequency, home, outdoors, going to void, during urinary urgency, nocturia). Severity of LUTSs were assessed by the Urinary Symptoms Profile (USP) Score and patient were classified as with or without urinary incontinence. Number of micturition by night were specifically asked. To take into account motor difficulties and fear of falling, other clinical evaluations were done. The impact of MS on walking was assessed by the 12-Item Multiple Sclerosis Walking Scale (MSWS12) questionnaire, the Expanded Disability Status Scale score, and by clinical test with the Time to be Ready to Void (TRV). Fear of falling was assessed by a simple question and with Falls Efficacy Scale-International (FES-I) Questionnaire.

The primary aim was to assess the relationship between severity of LUTSs and occurrence of falls during the past 3 months. The primary outcome was the importance of overactive bladder (OAB) symptoms with OAB USP score. The secondary outcomes were the existence of urinary incontinence, the warning time (defined as the time from the first sensation of urgency to voiding or incontinence), the importance of nocturia and the other scores of USP questionnaire (low stream and stress urinary incontinence).

The secondary aims were to look for the relationship between severity of LUTSs and occurrence of falls during the past year, and to assess the relationship between falls and the classical risk factors of falls.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* Multiple sclerosis (MS) diagnosis
* Lower urinary tract symptoms with or without treatment,
* Expanded Disability Status Scale score between 1 and 6.5

Exclusion Criteria:

* relapse of MS in the past month
* urinary tract infection the day of inclusion
* impossibility to complete the symptoms' questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting in a tertiary center in neuro-urology
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Number of falls in the past 3 months | 1 day
  Patients were asked about the number of falls in the past three months, and the circumstances in which they occurred (frequency, home, outdoors, going to void, during urinary urgency, nocturia)

SECONDARY OUTCOMES:
Number of falls in the past year | 1 day
  Patients were asked about the number of falls in the past year, and the circumstances in which they occurred (frequency, home, outdoors, going to void, during urinary urgency, nocturia)

OTHER OUTCOMES:
Correlation between number of falls in the past 3 months and in the past year and clinical datas and characteristics of the patient | 1 day
  The impact of MS on walking was assessed by the 12-Item Multiple Sclerosis Walking Scale (MSWS12) questionnaire, the EDSS score, and by clinical test with the Time to be Ready to Void (TRV). Fear of falling was assessed by a simple question and with Falls Efficacy Scale-International (FES-I) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PhD, Principal Investigator — Sorbonne Université, GRC 001, GREEN, AP-HP, Hôpital Tenon, Paris, France
Locations (1):
- department of Neuro-Urology, Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hentzen C, Villaume A, Turmel N, Chesnel C, Le Breton F, Haddad R, Amarenco G. Are falls in people with multiple sclerosis related to the severity of urinary disorders? Ann Phys Rehabil Med. 2021 Jul;64(4):101452. doi: 10.1016/j.rehab.2020.10.006. Epub 2020 Dec 5. PMID 33186783